CLINICAL TRIAL: NCT00185562
Title: A Pilot Trial of Adalimumab for the Treatment of Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-033
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2006-03-24 (Estimated); Status verified 2006-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
A 12 week trial of Adalimumab in subjects with active erosive inflammatory OA who have ahd an inadequate response to NSAID therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 45 or older, >/=2 tender and 2 swollen joints, inadequate response to NSAID therapy, hand radiographs with evidence of erosive changes, acceptable form of birth control

Exclusion Criteria:

* Autoimmune arthropathy, History of psoriasis, Previous TNF therapy, current use of any DMARD, evidence of TB, history of Hep C, B, or HIV

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-06; Study Completion 2006-01

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
20% ACR response

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Genovese, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States